CLINICAL TRIAL: NCT01549990
Title: A Comparison of Kidney Function After Nephrectomy in Living Donors Under Sevoflurane and Desflurane Anesthesia
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2012-0012
Record Dates: First submitted 2012-03-06; First posted 2012-03-09 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Nephrectomy,Kidney Donation
MeSH Terms: interventions — Sevoflurane; Desflurane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sevoflurane group: donors who went through donor nephrectomy under general anesthesia with sevoflurane
  Interventions: Drug: Sevoflurane
- desflurane group: donors who went through donor nephrectomy under general anesthesia with desflurane
  Interventions: Drug: desflurane

INTERVENTIONS:
Drug: Sevoflurane — maintenance of general anesthesia with sevoflurane
  Groups: Sevoflurane group
Drug: desflurane — maintenance of general anesthesia with desflurane
  Groups: desflurane group

SUMMARY:
Living-donor kidney transplantation has been considered as the best treatment for patients with end-stage renal disease (ESRD). Kidney donation from living donors has been performed widely under their noble humanity and a belief that donation would not harm the donor. Although the overall evidences proposed that living kidney donor have medical outcomes similar to those in general population, several reports have demonstrated the potential risks for development of hypertension, proteinuria, and ESRD. Thus, all efforts should be concentrated on ensuring their safety and preserving the function of their remained kidney during anesthesia maintenance.

Inhaled anesthetics have been frequently used for the induction and maintenance of general anesthesia. The metabolism of certain inhaled anesthetics can produce inorganic fluoride, which may be directly nephrotoxic through impairments of renal concentrating ability. The typical inhaled anesthetics commonly used nowadays are sevoflurane and desflurane. The defluorination of sevoflurane can results in increased serum inorganic fluoride ion concentrations, but any neprhotoxic effect of sevoflurane has not been proven yet in human. On the other hand, desflurane is extremely resistant to defluorination, and desflurane does not appear to be nephrotoxic.

The inhaled anesthetics which are currently used in general anesthesia have no clinical evidence of nephrotoxicity, but the possible risks cannot be excluded entirely, especially in the patients who one kidney is donated. The purpose of the current retrospective, single center study was to evaluate and compare postoperative renal function of living kidney donor after nephrectomy under sevoflurane or desflurane anesthesia, and make evidence-based recommendations of proper inhaled anesthetics for anesthesia of living kidney donor.

ELIGIBILITY:
Inclusion Criteria:

* donors who went through nephrectomy for kidney donation under general anesthesia with sevoflurane or desflurane

Exclusion Criteria:

* donors who went through nephrectomy for kidney donation under general anesthesia with other inhaled anesthetics except sevoflurane and desflurane

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From January 2006 through December 2011, donors who went through nephrectomy for kidney donation
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2012-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Postoperative renal function of living kidney donor after nephrectomy under sevoflurane or desflurane anesthesia | Participants will be followed for postoperative period, approximate 1 week through chart review.
  We collect laboratory data of the patients which were underwent at preoperative period and during postoperative periods. The laboratory data includes hemoglobin (Hb), hematocrit (Hct), platelet, prothrombin time (PT), albumin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), blood urea nitrogen (BUN), creatinine (Cr) and estimated glomerular filtration rate (eGFR) which was calculated by the Modification of Diet in Renal Disease (MDRD) formula with age, gender, race, and serum creatinine as variables.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Vats HS, Rayhill SC, Thomas CP. Early postnephrectomy donor renal function: laparoscopic versus open procedure. Transplantation. 2005 Mar 15;79(5):609-12. doi: 10.1097/01.tp.0000151662.84962.4e. PMID 15753853